CLINICAL TRIAL: NCT06375330
Title: Clinical Efficacy of Polynucleotides TMJ Injections Compared to Physiotherapy. A 3-months Randomized Clinical Trial.
Brief Title: Clinical Efficacy of Polynucleotides TMJ Injections Compared to Physiotherapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidoti & Tartaglia Srl (Other)
Responsible Party: Principal Investigator, Gianluca Tartaglia, Principal Investigator, Sidoti & Tartaglia Srl
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Poli.01
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: TMJ Disease; TMJ Pain
Keywords: polynucleotides; TMJ; VAS; Physiotherapy; Hyaluronic acid; Laterality
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 10 mg/ml Polynucleotides + 10 mg/ml Hyaluronic Acid in 2 mL prefilled syringe injections
  Interventions: Device: PoliArt
- Physiotherapy (No Intervention): Physiotherapy

INTERVENTIONS:
Device: PoliArt — PoliArt injections
  Arms: Treatment

SUMMARY:
The main objective of the present study is the evaluation of the clinical efficacy of the intra-articular administration of polynucleotides in association with hyaluronic acid in the improvement of the subjective and objective manifestations of arthrosis of the temporomandibular joint compared to normal clinical management which involves Physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients who signed the informed consent
* age >18;
* male and female sex;
* affected by temporomandibular arthrosis

Exclusion Criteria:

* Patients treated with painkillers and anti-inflammatories;
* patients suffering from rheumatoid arthritis with TMJ involvement;
* patients with a positive history of allergies to products of fish origin;
* patients suffering from alteration of the internal TMJ;
* patients suffering from mandibular condylar hyperplasia;
* patients suffering from myofascial pain syndrome;
* patients unable to express their consent for participation in the study;
* patients suffering from psychiatric and behavioral disorders;
* patients suffering from oncological and onco-haematological pathologies with compromised general clinical status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Maximum mouth opening | 3 months
  The primary objective is to evaluate the improvement of symptoms over time in terms of maximum mouth opening of patients (which in most cases is limited) treated with polynucleotides in association with hyaluronic acid compared to patients treated with physiotherapy exercises.

SECONDARY OUTCOMES:
Lateral movements improvements | 3 months
  Evaluation of the improvement of symptoms over time in terms of lateral movements in patients treated with polynucleotides in association with hyaluronic acid compared to patients treated with physiotherapy exercises.
  Lateral movements of the mandible were measured in millimeters as the distance between upper and lower midline at maximum lateral excursion; if the midlines were not centered at maximum intercuspation position, the midline shift in millimeters was added (if contralateral) or subtracted (if ipsilateral) to the recorded measurement.
Pain assessment | 3 months
  Evaluation of the reduction of pain in the two groups over time with Visual Analogue Scale (VAS). VAS score was recorded on a Likert scale ranging from 1 to 10, according to the subjective pain felt by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Tartaglia, MD, Principal Investigator — ORDINARY PROFESSOR Department of Biomedical, Surgical and Dental Sciences
Locations (1):
- UOC di Chirurgia Maxillo-Facciale e Odontostomatologia della Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No